CLINICAL TRIAL: NCT01769144
Title: Acticoat Absorbent and BCT Antimicrobial for STSG Donor Site on Thigh---A Randomised Controlled Trial
Brief Title: Acticoat Absorbent and BCT Antimicrobial for STSG Donor Site on Thigh
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Collaborators: Bio-medical Carbon Technology Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Kuei-Chang Hsu, Consultant Surgeon, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VGHKS12-CT9-09
Record Dates: First submitted 2013-01-10; First posted 2013-01-16 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-01

CONDITIONS: Wound Healing; Wound Infection; Pain; Pruritus; Cicatrix
Keywords: wound healing; wound infection; pain; pruritus; cicatrix; dressings; acticoat absorbent; BCT; KoCarbonAg
MeSH Terms: conditions — Wound Infection; Pain; Pruritus; Cicatrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acticoat Absorbent (Active Comparator): Acticoat Absorbent wound dressing
  Interventions: Device: Acticoat Absorbent
- BCT wound dressing (Experimental): wound dressing
  Interventions: Device: BCT

INTERVENTIONS:
Device: Acticoat Absorbent — wound dressing
  Arms: Acticoat Absorbent
Device: BCT — wound dressing
  Other Names: KoCarbonAg
  Arms: BCT wound dressing

SUMMARY:
This study aims to compare the effectiveness of two wound dressings, Acticoat Absorbent (AA) and BCT Antimicrobial (BCT) on Split Thickness Skin Graft (STSG) donor site.

DETAILED DESCRIPTION:
Seventy patients who undergo STSG procedure in Kaohsiung Veterans General Hospital will be recruited. Two donor sites of equal lengths and widths on the same thigh, which are at least 2 cm apart will be covered randomly with AA and BCT each. Wound healing rate and infection rate will be assessed at 7 and 14 days after surgery. Degrees of pain and itchiness will be assessed daily with Visual Analogue Scale for the first 7 post-operative days. Scar appearance will be assessed with Vancouver Scar Scale 1, 3 and 6 months post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* patients who need STSG, longer than 8 cm and wider than 5 cm, from their thighs

Exclusion Criteria:

* systemic steroid
* old scar on thigh
* systemic infection
* anticipated use of antibiotics for more than 24 hours after operation
* pregnancy
* previous chemotherapy within 3 months before operation
* anticipated chemotherapy within 3 months after operation
* not over 20 years old
* non-communicable
* burn area more than 20% total body surface area
* systemic auto-immune disease
* liver cirrhosis
* allergy to carbon fiber or alginate
* anticipated MRI study
* dry wound

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2013-01; Primary Completion 2013-07 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
wound healing rate | 7 days
  percentage of wound area that has healed at this time
wound infection rate | 7 days
wound healing rate | 14 days
  percentage of wound area that has healed at this time

SECONDARY OUTCOMES:
scar appearance | 1 month
pain and itchiness | 1day
scar appearance | 3 months
scar appearance | 6 months
pain and itchiness | 2 days
pain and itchiness | 3 days
pain and itchiness | 4 days
pain and itchiness | 5 days
pain and itchiness | 6 days
pain and itchiness | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Kuei-Chang Hsu, MD, Principal Investigator — Kaohsiung Veterans General Hospital.
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Background] Klasen HJ. Historical review of the use of silver in the treatment of burns. I. Early uses. Burns. 2000 Mar;26(2):117-30. doi: 10.1016/s0305-4179(99)00108-4. No abstract available. PMID 10716354
- [Background] Trop M, Novak M, Rodl S, Hellbom B, Kroell W, Goessler W. Silver-coated dressing acticoat caused raised liver enzymes and argyria-like symptoms in burn patient. J Trauma. 2006 Mar;60(3):648-52. doi: 10.1097/01.ta.0000208126.22089.b6. PMID 16531870
- [Background] Vlachou E, Chipp E, Shale E, Wilson YT, Papini R, Moiemen NS. The safety of nanocrystalline silver dressings on burns: a study of systemic silver absorption. Burns. 2007 Dec;33(8):979-85. doi: 10.1016/j.burns.2007.07.014. Epub 2007 Oct 23. PMID 17959313
- [Result] Tredget EE, Shankowsky HA, Groeneveld A, Burrell R. A matched-pair, randomized study evaluating the efficacy and safety of Acticoat silver-coated dressing for the treatment of burn wounds. J Burn Care Rehabil. 1998 Nov-Dec;19(6):531-7. doi: 10.1097/00004630-199811000-00013. PMID 9848045
- [Result] Argirova M, Hadjiski O, Victorova A. Acticoat versus Allevyn as a split-thickness skin graft donor-site dressing: a prospective comparative study. Ann Plast Surg. 2007 Oct;59(4):415-22. doi: 10.1097/SAP.0b013e3180312705. PMID 17901734
- [Result] Innes ME, Umraw N, Fish JS, Gomez M, Cartotto RC. The use of silver coated dressings on donor site wounds: a prospective, controlled matched pair study. Burns. 2001 Sep;27(6):621-7. doi: 10.1016/s0305-4179(01)00015-8. PMID 11525858
- [Result] Huang Y, Li X, Liao Z, Zhang G, Liu Q, Tang J, Peng Y, Liu X, Luo Q. A randomized comparative trial between Acticoat and SD-Ag in the treatment of residual burn wounds, including safety analysis. Burns. 2007 Mar;33(2):161-6. doi: 10.1016/j.burns.2006.06.020. Epub 2006 Dec 18. PMID 17175106
- [Result] Moiemen NS, Shale E, Drysdale KJ, Smith G, Wilson YT, Papini R. Acticoat dressings and major burns: systemic silver absorption. Burns. 2011 Feb;37(1):27-35. doi: 10.1016/j.burns.2010.09.006. Epub 2010 Oct 18. PMID 20961690